CLINICAL TRIAL: NCT04903977
Title: Clinical Performance and Safety of ONIRY Device in Detecting Obstetric Anal Sphincter Injuries Using Machine-learning-assisted Impedance Spectroscopy
Brief Title: Detection of Obstetric Anal Sphincter Injuries With ONIRY Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OASIS Diagnostics S.A. (Industry)
Collaborators: National Center for Research and Development, Poland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3/2/2020 AMD 02, Sep 16, 2022
Record Dates: First submitted 2021-05-17; First posted 2021-05-27 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Obstetric Anal Sphincter Injury; Delivery Complication; Obstetric Complication
Keywords: impedance spectroscopy; ONIRY; machine learning
MeSH Terms: interventions — Electrocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Impedance spectroscopy (Experimental): ONIRY examination
  Interventions: Diagnostic Test: Laboratory tests: blood and faeces tests; Diagnostic Test: Gynaecological and proctological examinations; Diagnostic Test: 3-D Endoanal Ultrasound; Device: ONIRY measurement; Diagnostic Test: High-resolution anorectal manometry; Diagnostic Test: ECG

INTERVENTIONS:
Diagnostic Test: Laboratory tests: blood and faeces tests — To be performed at V2
Diagnostic Test: Gynaecological and proctological examinations — To be performed at V1 (Examination with a gynaecological speculum, Bimanual examination, Rectal examination, and Anoscopy)
Diagnostic Test: 3-D Endoanal Ultrasound — To be performed at V1 (as a reference and for group assignment)
Device: ONIRY measurement — To be performed at V2 (the electrical impedance of anal sphincter muscles will be measured)
  Other Names: Impedance spectroscopy measurement
Diagnostic Test: High-resolution anorectal manometry — To be performed at V3
Diagnostic Test: ECG — To be performed at V1 and V2 (for safety reasons)

SUMMARY:
The main purpose of the study is to confirm the clinical performance and safety of impedance spectroscopy using the ONIRY device for the detection of anal sphincter injuries arising from vaginal deliveries.

The study group comprises 150 primiparous or multiparous women up to 8 weeks after the vaginal (spontaneous or assisted) delivery of singleton, live foetus, in any presentation, in gestational week 34 or more. The timeline for each subject in the study will be up to 5 weeks and will include 3 visits (V1-V3).

All participants will be divided into 3 groups: A, B, C. Group A - subjects with no perineal tear signs, Group B - subjects with grade 1 or 2 per OASIS classification, and Group C - subjects with grade 3 or 4).

The diagnostic performance will be evaluated in comparison to 3-D EUS (endoanal ultrasound) as a primary performance measure (primary endpoint).

DETAILED DESCRIPTION:
The main purpose of the study is to confirm the clinical performance and safety of impedance spectroscopy using the ONIRY device for the detection of anal sphincter injuries arising from vaginal deliveries. The whole study is divided into 2 parts. Part I is a clinical trial; after completion of Part I, an analytical classification model will be established (during Part II) based on data from pilot studies and Part I of the study. It will be then built into the ONIRY Meter as a machine-learning-based interpretation module; proposed for ultimate marketing authorisation.

Part I of the study will be prospective, multicentre, international. The study group comprises 150 primiparous or multiparous women up to 8 weeks after the vaginal (spontaneous or assisted) delivery of singleton, live foetus, in any presentation, in gestational week 34 or more. The timeline for each subject in the study will be up to 5 weeks and will include 3 visits (V1-V3).

After obtaining written consent, at the first study visit (V1) each patient will undergo a general physical examination, proctological and gynaecological examination, ECG recording, 3-D EUS (endoanal ultrasound, used as a reference and for the study group allocation) and once V1 visit is conducted 3 or more days after delivery Wexner score will be used to assess the clinical symptoms of faecal incontinence.

Based on the physical proctological examination and EUS at the V1 visit, all participants will be divided into 3 groups: A, B, C. Group A - subjects with no perineal tear signs, Group B - subjects with the presence of perineal skin injury or perineum injury involving crotch muscles but not involving anal sphincters (grade 1 or 2 per OASIS classification) and Group C - subjects with the presence of perineal injury involving anal sphincters (damage of the external anal sphincter thickness, damage to both the external and internal anal sphincters, or damage to the perineum, anal sphincteric complex and anal epithelium; grade 3-4).

On the visit V2 performed on the same day as V1 or scheduled up to 7 days after the V1, after the final verification of inclusion/exclusion criteria, blood samples for laboratory tests and stool samples for calprotectin concentration assessment will be collected, ONIRY recording will be made, 10 minutes after the end of the impedance measurement 12-lead ECG recording will also be performed in each patient.

On the third visit (V3) 1-28 days after visit V2, high-resolution Anorectal Manometry will be conducted.

No control group is planned. However, study participants will be controls for themselves (test and reference diagnostic methods will be applied and evaluated in each subject).

In Part I of the study, the ONIRY system will provide only preliminary interpretations of the impedance measurements based on models established from the data collected during Pilot Studies No. 1/1/2018 (NCT03769792) and No. 2/1/2019 (NCT04181840). The web-based app will be used to provide the interpretations.

ELIGIBILITY:
Inclusion Criteria:

1. Women between 18 and 49 years old;
2. Primiparous or multiparous;
3. Since the first moments up to 8 weeks after vaginal delivery (including spontaneous and assisted):

   1. of singleton, live foetus,
   2. in any presentation,
   3. in gestational week 34 or more.
4. For group A:

   1. no clinical signs of any degree perineal tear
   2. no clinical signs or symptoms of any damage involving anal sphincters;
   3. presence of not more than 1 of following OASIS risk factors related to the last delivery: prolonged second phase of delivery, foetal shoulder dystocia, birth weight of the neonate >4kg, induction of delivery using oxytocin, or head circumference of the neonate ≥34 cm
5. For groups B and C:

   1. clinically confirmed 1 or 2-degree perineal tear (including episiotomy and uncontrolled crotch rupture) occurred at the last delivery (for group B);
   2. clinically identified 3 or 4-degree perineal tear (damage involving anal sphincters) occurred at the last delivery (regardless of primary repair) (for group C);
6. Signed informed consent form (no proxy or witnessed consent allowed).

Exclusion Criteria:

1. Any acute, uncontrolled disease (except for haemorrhoidal disease)
2. Chronic diseases not treated or not stable on treatment;
3. Symptoms of faecal incontinence due to a disease other than diagnosed or suspected OASIS;
4. Previous surgery for OASIS (primary or secondary), faecal incontinence or anal prolapse, except for a primary repair of anal sphincter damage performed after the last delivery (allowed);
5. Any surgery in perineal or rectal area, including surgery for OASIS, planned for the study period
6. Presence of inflammatory bowel diseases during exacerbation phase;
7. Any treatment during last 12 months for severe, progressive, uncontrolled cardiological, pulmonary, nephrology, contagious or psychiatric illness that could increase subject's risk due to participation in the study,
8. Disease other than OASIS so far undiagnosed and reported during the visit V1 or within 7 days prior to it;
9. Present or suspected malignancy or previous oncological treatment in the last 5 years;
10. Implanted cardiac stimulator or cardioverter-defibrillator;
11. Clinically significant cardiac arrhythmias observed in ECG examination or reported in history for the last 12 months;
12. Fever (>37°C) at enrolment;
13. History of major surgery in perineal or rectal area (other than for OASIS) or severe trauma of perineum or rectum.
14. Use, or need for use, of an anal suppository or other anally administered drug, or cosmetic for the perianal area, within 12 hours prior to impedance spectroscopy examination (visit V2).
15. Positive pregnancy test (only for subjects recruited ≥4 weeks after delivery with no lactation at V1 visit; however, subjects with a positive pregnancy test may be enrolled as long as gynaecologic ultrasound performed at V1 visit shows no signs of a new pregnancy, no sings suggestive of placental tissue remaining in utero, or other abnormality of the uterus).

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 152 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2022-12-08 (Actual)

PRIMARY OUTCOMES:
Diagnostic Outcome in Clinically-evaluable (CE) Population with 3-D EUS used as the reference diagnostic method | Up to 9 weeks post-partum
  The Diagnostic Outcome defined as Diagnostic Success, Diagnostic Failure or Indeterminate, will be programmatically determined for each subject:
  a. Diagnostic Success: i. occurrence of an anal sphincter injury; or ii. absence of an anal sphincter injury; confirmed consistently by ONIRY and the reference diagnostic method (True Positive, TP, or True Negative, TN, respectively); b. Diagnostic Failure: i. occurrence of anal sphincter injury detected by ONIRY and absence of anal sphincter injury found out using the reference diagnostic method (False Positive, FP) or ii. absence of anal sphincter injury by ONIRY and occurrence of anal sphincter injury found out using the reference diagnostic method (False Negative, FN); c. Diagnostic Indeterminate - all cases in which no ONIRY or reference diagnostic method result is available or interpretable.

SECONDARY OUTCOMES:
Diagnostic Outcome in CE Population with physical rectal examination used as the reference diagnostic method | Up to 9 weeks post-partum
  The Diagnostic Outcome defined as Diagnostic Success, Diagnostic Failure or Indeterminate, will be programmatically determined for each subject:
  a. Diagnostic Success: i. occurrence of an anal sphincter injury; or ii. absence of an anal sphincter injury; confirmed consistently by ONIRY and the reference diagnostic method (True Positive, TP, or True Negative, TN, respectively); b. Diagnostic Failure: i. occurrence of anal sphincter injury detected by ONIRY and absence of anal sphincter injury found out using the reference diagnostic method (False Positive, FP) or ii. absence of anal sphincter injury by ONIRY and occurrence of anal sphincter injury found out using the reference diagnostic method (False Negative, FN); c. Diagnostic Indeterminate - all cases in which no ONIRY or reference diagnostic method result is available or interpretable.
Diagnostic Outcome in CE Population with high-resolution anorectal manometry used as the reference diagnostic method | Up to 13 weeks post-partum
  The Diagnostic Outcome defined as Diagnostic Success, Diagnostic Failure or Indeterminate, will be programmatically determined for each subject:
  a. Diagnostic Success: i. occurrence of an anal sphincter injury; or ii. absence of an anal sphincter injury; confirmed consistently by ONIRY and the reference diagnostic method (True Positive, TP, or True Negative, TN, respectively); b. Diagnostic Failure: i. occurrence of anal sphincter injury detected by ONIRY and absence of anal sphincter injury found out using the reference diagnostic method (False Positive, FP) or ii. absence of anal sphincter injury by ONIRY and occurrence of anal sphincter injury found out using the reference diagnostic method (False Negative, FN); c. Diagnostic Indeterminate - all cases in which no ONIRY or reference diagnostic method result is available or interpretable.
Occurrence of AEs in Safety Population | Up to 13 weeks post-partum
  Assessment of the safety of the device

OTHER OUTCOMES:
Correlation of faecal incontinence symptoms, assessed using Wexner score, with ONIRY, 3-D EUS, physical rectal examination, and high-resolution anorectal manometry results in Safety Population | Up to 13 weeks post-partum
  Exploratory endpoint #1
Diagnostic Outcome in CE Population with 3-D EUS used as the reference diagnostic method utilising the classification of anal sphincter injuries according to Starck | Up to 13 weeks post-partum
  Exploratory endpoint #2
Diagnostic Outcome in CE Population with 3-D EUS used as the reference diagnostic method utilising the classification of anal sphincter injuries according to Norderval | Up to 13 weeks post-partum
  Exploratory endpoint #3

CONTACTS AND LOCATIONS:
Locations (5):
- Czechia (2):
  - Fakultni nemocnice, Brno
  - Ustav pro peci o matku a dite, Prague
- FEMINITY Praktyka Lekarska dr Małgorzata Uchman-Musielak, Warsaw, Poland
- Gynekologicko-pôrodnícka klinika Nemocnica AGEL Košice-Šaca a.s., Košice, Košice Region, Slovakia
- Complejo Asistencial Universitario de Leon, León, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor's website — https://www.oasis-diagnostics.com